CLINICAL TRIAL: NCT00226044
Title: Rectal and Oral Omeprazole Treatment of Gastroesophageal Reflux in Infants With Esophageal Atresia or Congenital Diaphragmatic Hernia; A Pharmacodynamic and Pharmacokinetic Study.
Brief Title: Rectal and Oral Omeprazole Treatment of Reflux Disease in Infants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTC-001
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Gastroesophageal Reflux; Esophageal Atresia; Hernia, Diaphragmatic
Keywords: Omeprazole, suppository, infants
MeSH Terms: conditions — Gastroesophageal Reflux; Esophageal Atresia; Hernia, Diaphragmatic

STUDY DESIGN:
Intervention Model Description: This study was an open-label randomized intervention trial to study the efficacy of a single oral or rectal administered omeprazole dose of 1 mg/kg in infants with GERD due to EA or CDH.

ARMS (2):
- Oral omeprazole (No Intervention): Standard of care: A single dose of 1 mg/kg orally administered omeprazole.
- Rectal omeprazole (Active Comparator): A single dose of 1 mg/kg rectally administered omeprazole.
  Interventions: Drug: Omeprazole rectally 1mg/kg

INTERVENTIONS:
Drug: Omeprazole rectally 1mg/kg — A single dose of 1 mg/kg rectally administered omeprazole.
  Arms: Rectal omeprazole

SUMMARY:
The purpose of this study is to compare the efficacy of oral and rectal omeprazole treatment in infants with gastroesophageal reflux due to esophageal atresia or congenital diaphragmatic hernia.

DETAILED DESCRIPTION:
Omeprazole is a highly effective drug for the treatment of gastroesophageal reflux disease (GERD) in infants. Infants, aged 0-12 months, require a non-standard dose of omeprazole. Due to this fact extemporaneous formulations of omeprazole are administered to these infants. The oral bioavailability of omeprazole in nonproprietary formulations may be unpredictable and produce variable degrees of drug exposure. The dose range for GERD management in pediatric studies using omeprazole is 0.3 - 3.5 mg/kg/day.

Dosing information, aged-specific pharmacodynamic and pharmacokinetic data are not available in infants, aged 0-12 months. Two adult studies at healthy volunteers suggest that an omeprazole suppository is an effective dosage form.This study is designed to evaluate and to compare the efficacy, the pharmacodynamics and the pharmacokinetics of oral and rectal omeprazole treatment in infants with gastroesophageal reflux disease.

ELIGIBILITY:
Infants were eligible for the study if they were:

* 6-12 weeks postnatal age
* weighed more than 3 kg
* were after surgical repair for EA or CDH
* showed clinical GERD
* were to undergo the 48 hour pH measurements.

Infants were excluded if they were:

* allergic to omeprazole
* participated in other interventional trials
* used medications known to interact with omeprazole.

Ages: 6 Weeks to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy | 24 hour
  Primary: percentage of infants for which omeprazole was effective according to predefined criteria for 24 hour intraesophageal pH.

SECONDARY OUTCOMES:
Intragastric pH | 24 hours
  Secondary: outcomes were the percentage of time gastric pH was <3 and <4
Maximum plasma concentration (Cmax) | 8 hours
  The maximal concentration of OME, OH-OME and OME-S in plasma (Cmax)
Time to reach Cmax (Tmax) | 8 hours
  time to reach Cmax (Tmax)
Area under the curve (AUC) | 8 hours
  The AUC from time zero to the last sampling time point (AUC0-t)

CONTACTS AND LOCATIONS:
Overall Officials: S.N. de Wildt, Prof. Dr., Study Director — Erasmus Medical Center
Locations (1):
- Erasmus Medical center, Rotterdam, Netherlands

REFERENCES:
- [Derived] Bestebreurtje P, de Koning BAE, Roeleveld N, Knibbe CAJ, Tibboel D, van Groen B, van de Ven CP, Plotz FB, de Wildt SN. Rectal Omeprazole in Infants With Gastroesophageal Reflux Disease: A Randomized Pilot Trial. Eur J Drug Metab Pharmacokinet. 2020 Oct;45(5):635-643. doi: 10.1007/s13318-020-00630-8. PMID 32594305